CLINICAL TRIAL: NCT03918252
Title: Neoadjuvant Immune Checkpoint Blockade in Resectable Malignant Pleural Mesothelioma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: J1932; IRB00203283 (Other: JHM IRB)
Record Dates: First submitted 2019-04-15; First posted 2019-04-17 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Mesothelioma
Keywords: malignant; resectable
MeSH Terms: conditions — Mesothelioma | interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A Nivolumab Only (Experimental): Receive preoperative nivolumab, 240mg IV, on Day -42, -28 and Day -14 (+/- two days for each timepoint) prior to planned surgery on Day 0 (to allow for scheduling surgery may take place between Day -3 and Day +10).
  Interventions: Drug: Nivolumab Injection
- Arm B Nivolumab + Ipilimumab (Experimental): Receive preoperative nivolumab, 3mg/kg IV, on Day -42, -28 and Day -14 (+/- two days for each timepoint) + ipilimumab 1mg/kg IV on Day -42 prior to planned surgery on Day 0 (to allow for scheduling surgery may take place between Day -3 and Day +10).
  Interventions: Drug: Nivolumab Injection; Drug: Ipilimumab Injection

INTERVENTIONS:
Drug: Nivolumab Injection — Receive preoperative nivolumab, 240mg IV, on Day -42, -28 and Day -14 (+/- two days for each timepoint) prior to planned surgery on Day 0 (to allow for scheduling surgery may take place between Day -3 and Day +10).
  Other Names: Optivo
Drug: Ipilimumab Injection — Receive preoperative nivolumab, 3mg/kg IV, on Day -42, -28 and Day -14 (+/- two days for each timepoint) + ipilimumab 1mg/kg IV on Day -42 prior to planned surgery on Day 0 (to allow for scheduling surgery may take place between Day -3 and Day +10).
  Other Names: Yervoy
  Arms: Arm B Nivolumab + Ipilimumab

SUMMARY:
The proposed study will evaluate the safety and feasibility of neoadjuvant nivolumab +/- ipilimumab in resectable MPM. In addition, maintenance nivolumab will be administered for 1 year following completion of standard bi-/tri-modality therapy.

DETAILED DESCRIPTION:
For Arm A 15 patients with resectable MPM will be enrolled and receive preoperative nivolumab, 240mg IV, on Day -42, -28 and Day -14 (+/- two days for each timepoint) prior to planned surgery on Day 0 (to allow for scheduling surgery may take place between Day -3 and Day +10).

Subsequent to full accrual to Arm A, 15 patients with resectable MPM will be enrolled and receive preoperative nivolumab, 3mg/kg IV, on Day -42, -28 and Day -14 (+/- two days for each timepoint) + ipilimumab 1mg/kg IV on Day -42 prior to planned surgery on Day 0 (to allow for scheduling surgery may take place between Day -3 and Day +10).

ELIGIBILITY:
Inclusion Criteria:

* Men and women ≥ 18 years old
* Primary tumor amenable to safe research biopsy. A tumor biopsy is required for study entry.
* Histology proven epithelial or biphasic MPM

  * Diagnostic core biopsy specimens must be reviewed by faculty pathologist at SKCC, MDACC, or UMGCCC.
  * Either a formalin fixed paraffin block that has been confirmed by a pathologist to contain tumor or a minimum of twenty 5-micron tissue sections (slides) of tumor biopsy sample must be available for biomarker evaluation (study pathologist must review for adequacy of sampling). This can be obtained from archived tissues if adequate, or from a new biopsy as needed.
* Stage I-III and deemed to be potentially surgically resectable as assessed by faculty surgeon at SKCC, MDACC, or UMGCCC
* ECOG performance status 0-1
* Adequate organ function as follows:

  * Leukocytes ≥ 2,000/mm3
  * Absolute neutrophil count (ANC) ≥ 1000/mm3
  * Platelet count ≥ 100,000/mm3
  * Hemoglobin ≥ 9 g/Dl
  * Creatinine ≤ 1.5 x ULN or creatinine clearance (CrCl) ≥40 mL/min (if using the Cockcroft-Gault formula below):

Female CrCl = (140 - age in years) x weight in kg x 0.85 72 x serum creatinine in mg/dL

Male CrCl = (140 - age in years) x weight in kg x 1.00 72 x serum creatinine in mg/dL

* Total Bilirubin ≤ 1.5 x institutional ULN (except subjects with Gilbert Syndrome, who can have total bilirubin < 3.0 mg/dL)
* AST(SGOT), ALT(SGPT), and alkaline phosphatase ≤ 3 times the institutional upper limit of normal
* Subjects must have adequate lung function to permit surgical resection determined by pre-enrollment pulmonary function tests to include DLCO

  * The effects of nivolumab on the developing human fetus are unknown. For this reason, women of child-bearing potential (WOCBP) and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation and for up to 23 weeks after the last dose of nivolumab. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Sexually active fertile men must use effective barrier birth control if their partners are WOCBP for up to 31 weeks after the last dose of nivolumab. WOCBP must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within two weeks of registration. Women must not be breastfeeding.
  * Patient understands the study regimen, its requirements, risks and discomforts and is able and willing to sign the informed consent form. Voluntary signed and dated IRB/IEC approved written informed consent form in accordance with regulatory and institutional guidelines must be obtained before the performance of any protocol related procedures that are not part of normal patient care. Subjects must be competent to report AEs, understand the drug dosing schedule and use of medications to control AEs.

Exclusion Criteria:

* Stage I-III disease but deemed to be unresectable, a poor surgical candidate, or unfit for study therapy as assessed by study investigators
* Pure sarcomatoid histology
* Subjects are excluded if they have an active, known or suspected autoimmune disease. Subjects are permitted to enroll if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger.
* Subjects are excluded if they have a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease. As there is potential for hepatic toxicity with nivolumab or nivolumab/ipilimumab combinations, drugs with a predisposition to hepatotoxicity should be used with caution in patients treated with nivolumab-containing regimen.
* Administration of chemotherapy or any other cancer therapy in the pre-operative period.
* Subjects with active concurrent malignancies are excluded i.e. cancers other than MPM (except non-melanoma skin cancers, cervical dysplasia, and in situ cancers of bladder, stomach, breast, colon and cervix).
* Subjects with a history of symptomatic interstitial lung disease.
* Active systemic infection requiring therapy, as well as positive tests for hepatitis B surface antigen or hepatitis C antibody.
* Known positive history or positive test for human immunodeficiency virus or Acquired Immunodeficiency Syndrome (AIDS).
* History of allergy to study drug components.
* Women who are pregnant or nursing.
* Men with female partners (WOCBP) that are unwilling to use contraception
* Prior therapy with an anti-PD1, anti-PD-L1, anti-PD-L2, or anti-CTLA-4 antibody (or any other antibody targeting T-cell co-regulatory pathways).
* History of any other condition that may require the initiation of anti-tumor necrosis factor alpha (TNFα) therapies or other immunosuppressant medications during the study
* Underlying medical conditions that, in the Investigator's opinion, will make the administration of study drug hazardous or obscure the interpretation of toxicity or adverse events.
* Prisoners or subjects who are involuntarily incarcerated or compulsorily detained for treatment of either a psychiatric or physical (e.g. infectious disease) illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-10-02 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Safety Profile of neoadjuvant nivolumab +/- ipilimumab in patients with resectable malignant pleural mesothelioma (MPM) with grade III/IV adverse events defined by CTCAE v5.0 | up to 5 years
  Number of participants with grade III/IV adverse events defined by CTCAE v5.0, occurring within 100 days of last study drug administration or 30 days post-surgery (whichever is longer).
Feasibility of neoadjuvant nivolumab +/- ipilimumab in patients with resectable MPM who complete of neoadjuvant treatment and proceed to surgery | up to 5 years
  Feasibility as measured by the number of participants who complete of neoadjuvant treatment with nivolumab +/- ipilimumab and proceed to surgery without extended treatment-related delay (>24 days from preplanned surgery date).

SECONDARY OUTCOMES:
Pathological Response to neoadjuvant nivolumab +/- ipilimumab in resected tumor and lymph nodes in patients with resectable MPM defined as ≤10% residual viable tumor cells and pathologic complete response | 5 years
  Number of participants with pathologic response, defined as ≤10% residual viable tumor cells in the resection specimen, and pathologic complete response (no residual viable tumor cells in the resection specimen).
Radiographic Response to neoadjuvant nivolumab +/- ipilimumab utilizing RECIST 1.1 | 5 years
  Number of participants with radiographic response as determined utilizing RECIST 1.1, modified RECIST for pleural tumors, and change in FDG avidity on PET/CT pre- and post-treatment.
Toxicity as assessed by number of participants experienced grade III/IV adverse events as defined by CTCAE v5.0 within 100 days of last study drug administration | up to 100 days post-intervention
  Toxicity as assessed by number of participants experienced grade III/IV adverse events as defined by CTCAE v5.0 within 100 days of last study drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Julie Brahmer, MD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (3):
- United States (3):
  - Greenebaum Comprehensive Cancer Center University of Maryland School of Medicine, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland
  - University of Texas M.D. Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tsao AS, Wistuba I, Roth JA, Kindler HL. Malignant pleural mesothelioma. J Clin Oncol. 2009 Apr 20;27(12):2081-90. doi: 10.1200/JCO.2008.19.8523. Epub 2009 Mar 2. PMID 19255316
- [Background] Mazurek JM, Syamlal G, Wood JM, Hendricks SA, Weston A. Malignant Mesothelioma Mortality - United States, 1999-2015. MMWR Morb Mortal Wkly Rep. 2017 Mar 3;66(8):214-218. doi: 10.15585/mmwr.mm6608a3. PMID 28253224
- [Background] Patil NS, Righi L, Koeppen H, Zou W, Izzo S, Grosso F, Libener R, Loiacono M, Monica V, Buttigliero C, Novello S, Hegde PS, Papotti M, Kowanetz M, Scagliotti GV. Molecular and Histopathological Characterization of the Tumor Immune Microenvironment in Advanced Stage of Malignant Pleural Mesothelioma. J Thorac Oncol. 2018 Jan;13(1):124-133. doi: 10.1016/j.jtho.2017.09.1968. Epub 2017 Oct 24. PMID 29079455
- [Background] Butchart EG, Ashcroft T, Barnsley WC, Holden MP. Pleuropneumonectomy in the management of diffuse malignant mesothelioma of the pleura. Experience with 29 patients. Thorax. 1976 Feb;31(1):15-24. doi: 10.1136/thx.31.1.15. PMID 1257933
- [Background] Weder W, Stahel RA, Bernhard J, Bodis S, Vogt P, Ballabeni P, Lardinois D, Betticher D, Schmid R, Stupp R, Ris HB, Jermann M, Mingrone W, Roth AD, Spiliopoulos A; Swiss Group for Clinical Cancer Research. Multicenter trial of neo-adjuvant chemotherapy followed by extrapleural pneumonectomy in malignant pleural mesothelioma. Ann Oncol. 2007 Jul;18(7):1196-202. doi: 10.1093/annonc/mdm093. Epub 2007 Apr 11. PMID 17429100
- [Background] Krug LM, Pass HI, Rusch VW, Kindler HL, Sugarbaker DJ, Rosenzweig KE, Flores R, Friedberg JS, Pisters K, Monberg M, Obasaju CK, Vogelzang NJ. Multicenter phase II trial of neoadjuvant pemetrexed plus cisplatin followed by extrapleural pneumonectomy and radiation for malignant pleural mesothelioma. J Clin Oncol. 2009 Jun 20;27(18):3007-13. doi: 10.1200/JCO.2008.20.3943. Epub 2009 Apr 13. PMID 19364962
- [Background] Treasure T, Lang-Lazdunski L, Waller D, Bliss JM, Tan C, Entwisle J, Snee M, O'Brien M, Thomas G, Senan S, O'Byrne K, Kilburn LS, Spicer J, Landau D, Edwards J, Coombes G, Darlison L, Peto J; MARS trialists. Extra-pleural pneumonectomy versus no extra-pleural pneumonectomy for patients with malignant pleural mesothelioma: clinical outcomes of the Mesothelioma and Radical Surgery (MARS) randomised feasibility study. Lancet Oncol. 2011 Aug;12(8):763-72. doi: 10.1016/S1470-2045(11)70149-8. Epub 2011 Jun 30. PMID 21723781
- [Background] Dunn GP, Bruce AT, Ikeda H, Old LJ, Schreiber RD. Cancer immunoediting: from immunosurveillance to tumor escape. Nat Immunol. 2002 Nov;3(11):991-8. doi: 10.1038/ni1102-991. PMID 12407406
- [Background] Retsas S, Priestman TJ, Newton KA, Westbury G. Evaluation of human lymphoblastoid interferon in advanced malignant melanoma. Cancer. 1983 Jan 15;51(2):273-6. doi: 10.1002/1097-0142(19830115)51:23.0.co;2-k. PMID 6821816
- [Background] West WH, Tauer KW, Yannelli JR, Marshall GD, Orr DW, Thurman GB, Oldham RK. Constant-infusion recombinant interleukin-2 in adoptive immunotherapy of advanced cancer. N Engl J Med. 1987 Apr 9;316(15):898-905. doi: 10.1056/NEJM198704093161502. PMID 3493433
- [Background] Tao MH, Levy R. Idiotype/granulocyte-macrophage colony-stimulating factor fusion protein as a vaccine for B-cell lymphoma. Nature. 1993 Apr 22;362(6422):755-8. doi: 10.1038/362755a0. PMID 8469286
- [Background] Phan GQ, Attia P, Steinberg SM, White DE, Rosenberg SA. Factors associated with response to high-dose interleukin-2 in patients with metastatic melanoma. J Clin Oncol. 2001 Aug 1;19(15):3477-82. doi: 10.1200/JCO.2001.19.15.3477. PMID 11481353
- [Background] Joseph RW, Sullivan RJ, Harrell R, Stemke-Hale K, Panka D, Manoukian G, Percy A, Bassett RL, Ng CS, Radvanyi L, Hwu P, Atkins MB, Davies MA. Correlation of NRAS mutations with clinical response to high-dose IL-2 in patients with advanced melanoma. J Immunother. 2012 Jan;35(1):66-72. doi: 10.1097/CJI.0b013e3182372636. PMID 22130161
- [Background] Krummel MF, Allison JP. CD28 and CTLA-4 have opposing effects on the response of T cells to stimulation. J Exp Med. 1995 Aug 1;182(2):459-65. doi: 10.1084/jem.182.2.459. PMID 7543139
- [Background] Leach DR, Krummel MF, Allison JP. Enhancement of antitumor immunity by CTLA-4 blockade. Science. 1996 Mar 22;271(5256):1734-6. doi: 10.1126/science.271.5256.1734. PMID 8596936
- [Background] Hodi FS, O'Day SJ, McDermott DF, Weber RW, Sosman JA, Haanen JB, Gonzalez R, Robert C, Schadendorf D, Hassel JC, Akerley W, van den Eertwegh AJ, Lutzky J, Lorigan P, Vaubel JM, Linette GP, Hogg D, Ottensmeier CH, Lebbe C, Peschel C, Quirt I, Clark JI, Wolchok JD, Weber JS, Tian J, Yellin MJ, Nichol GM, Hoos A, Urba WJ. Improved survival with ipilimumab in patients with metastatic melanoma. N Engl J Med. 2010 Aug 19;363(8):711-23. doi: 10.1056/NEJMoa1003466. Epub 2010 Jun 5. PMID 20525992
- [Background] Eggermont AM, Chiarion-Sileni V, Grob JJ, Dummer R, Wolchok JD, Schmidt H, Hamid O, Robert C, Ascierto PA, Richards JM, Lebbe C, Ferraresi V, Smylie M, Weber JS, Maio M, Bastholt L, Mortier L, Thomas L, Tahir S, Hauschild A, Hassel JC, Hodi FS, Taitt C, de Pril V, de Schaetzen G, Suciu S, Testori A. Prolonged Survival in Stage III Melanoma with Ipilimumab Adjuvant Therapy. N Engl J Med. 2016 Nov 10;375(19):1845-1855. doi: 10.1056/NEJMoa1611299. Epub 2016 Oct 7. PMID 27717298
- [Background] Zhang X, Schwartz JC, Guo X, Bhatia S, Cao E, Lorenz M, Cammer M, Chen L, Zhang ZY, Edidin MA, Nathenson SG, Almo SC. Structural and functional analysis of the costimulatory receptor programmed death-1. Immunity. 2004 Mar;20(3):337-47. doi: 10.1016/s1074-7613(04)00051-2. PMID 15030777
- [Background] Nishimura H, Honjo T. PD-1: an inhibitory immunoreceptor involved in peripheral tolerance. Trends Immunol. 2001 May;22(5):265-8. doi: 10.1016/s1471-4906(01)01888-9. PMID 11323285
- [Background] Freeman GJ, Long AJ, Iwai Y, Bourque K, Chernova T, Nishimura H, Fitz LJ, Malenkovich N, Okazaki T, Byrne MC, Horton HF, Fouser L, Carter L, Ling V, Bowman MR, Carreno BM, Collins M, Wood CR, Honjo T. Engagement of the PD-1 immunoinhibitory receptor by a novel B7 family member leads to negative regulation of lymphocyte activation. J Exp Med. 2000 Oct 2;192(7):1027-34. doi: 10.1084/jem.192.7.1027. PMID 11015443
- [Background] Latchman Y, Wood CR, Chernova T, Chaudhary D, Borde M, Chernova I, Iwai Y, Long AJ, Brown JA, Nunes R, Greenfield EA, Bourque K, Boussiotis VA, Carter LL, Carreno BM, Malenkovich N, Nishimura H, Okazaki T, Honjo T, Sharpe AH, Freeman GJ. PD-L2 is a second ligand for PD-1 and inhibits T cell activation. Nat Immunol. 2001 Mar;2(3):261-8. doi: 10.1038/85330. PMID 11224527
- [Background] Carter L, Fouser LA, Jussif J, Fitz L, Deng B, Wood CR, Collins M, Honjo T, Freeman GJ, Carreno BM. PD-1:PD-L inhibitory pathway affects both CD4(+) and CD8(+) T cells and is overcome by IL-2. Eur J Immunol. 2002 Mar;32(3):634-43. doi: 10.1002/1521-4141(200203)32:33.0.CO;2-9. PMID 11857337
- [Background] Chemnitz JM, Parry RV, Nichols KE, June CH, Riley JL. SHP-1 and SHP-2 associate with immunoreceptor tyrosine-based switch motif of programmed death 1 upon primary human T cell stimulation, but only receptor ligation prevents T cell activation. J Immunol. 2004 Jul 15;173(2):945-54. doi: 10.4049/jimmunol.173.2.945. PMID 15240681
- [Background] Sheppard KA, Fitz LJ, Lee JM, Benander C, George JA, Wooters J, Qiu Y, Jussif JM, Carter LL, Wood CR, Chaudhary D. PD-1 inhibits T-cell receptor induced phosphorylation of the ZAP70/CD3zeta signalosome and downstream signaling to PKCtheta. FEBS Lett. 2004 Sep 10;574(1-3):37-41. doi: 10.1016/j.febslet.2004.07.083. PMID 15358536
- [Background] Nishimura H, Nose M, Hiai H, Minato N, Honjo T. Development of lupus-like autoimmune diseases by disruption of the PD-1 gene encoding an ITIM motif-carrying immunoreceptor. Immunity. 1999 Aug;11(2):141-51. doi: 10.1016/s1074-7613(00)80089-8. PMID 10485649
- [Background] Nishimura H, Okazaki T, Tanaka Y, Nakatani K, Hara M, Matsumori A, Sasayama S, Mizoguchi A, Hiai H, Minato N, Honjo T. Autoimmune dilated cardiomyopathy in PD-1 receptor-deficient mice. Science. 2001 Jan 12;291(5502):319-22. doi: 10.1126/science.291.5502.319. PMID 11209085
- [Background] Wang J, Yoshida T, Nakaki F, Hiai H, Okazaki T, Honjo T. Establishment of NOD-Pdcd1-/- mice as an efficient animal model of type I diabetes. Proc Natl Acad Sci U S A. 2005 Aug 16;102(33):11823-8. doi: 10.1073/pnas.0505497102. Epub 2005 Aug 8. PMID 16087865
- [Background] Okazaki T, Tanaka Y, Nishio R, Mitsuiye T, Mizoguchi A, Wang J, Ishida M, Hiai H, Matsumori A, Minato N, Honjo T. Autoantibodies against cardiac troponin I are responsible for dilated cardiomyopathy in PD-1-deficient mice. Nat Med. 2003 Dec;9(12):1477-83. doi: 10.1038/nm955. Epub 2003 Nov 2. PMID 14595408
- [Background] Konishi J, Yamazaki K, Azuma M, Kinoshita I, Dosaka-Akita H, Nishimura M. B7-H1 expression on non-small cell lung cancer cells and its relationship with tumor-infiltrating lymphocytes and their PD-1 expression. Clin Cancer Res. 2004 Aug 1;10(15):5094-100. doi: 10.1158/1078-0432.CCR-04-0428. PMID 15297412
- [Background] Thompson RH, Gillett MD, Cheville JC, Lohse CM, Dong H, Webster WS, Krejci KG, Lobo JR, Sengupta S, Chen L, Zincke H, Blute ML, Strome SE, Leibovich BC, Kwon ED. Costimulatory B7-H1 in renal cell carcinoma patients: Indicator of tumor aggressiveness and potential therapeutic target. Proc Natl Acad Sci U S A. 2004 Dec 7;101(49):17174-9. doi: 10.1073/pnas.0406351101. Epub 2004 Nov 29. PMID 15569934
- [Background] Ohigashi Y, Sho M, Yamada Y, Tsurui Y, Hamada K, Ikeda N, Mizuno T, Yoriki R, Kashizuka H, Yane K, Tsushima F, Otsuki N, Yagita H, Azuma M, Nakajima Y. Clinical significance of programmed death-1 ligand-1 and programmed death-1 ligand-2 expression in human esophageal cancer. Clin Cancer Res. 2005 Apr 15;11(8):2947-53. doi: 10.1158/1078-0432.CCR-04-1469. PMID 15837746
- [Background] Tsushima F, Tanaka K, Otsuki N, Youngnak P, Iwai H, Omura K, Azuma M. Predominant expression of B7-H1 and its immunoregulatory roles in oral squamous cell carcinoma. Oral Oncol. 2006 Mar;42(3):268-74. doi: 10.1016/j.oraloncology.2005.07.013. Epub 2005 Nov 3. PMID 16271509
- [Background] Thompson RH, Webster WS, Cheville JC, Lohse CM, Dong H, Leibovich BC, Kuntz SM, Sengupta S, Kwon ED, Blute ML. B7-H1 glycoprotein blockade: a novel strategy to enhance immunotherapy in patients with renal cell carcinoma. Urology. 2005 Nov;66(5 Suppl):10-4. doi: 10.1016/j.urology.2005.06.010. PMID 16194701
- [Background] Thompson RH, Gillett MD, Cheville JC, Lohse CM, Dong H, Webster WS, Chen L, Zincke H, Blute ML, Leibovich BC, Kwon ED. Costimulatory molecule B7-H1 in primary and metastatic clear cell renal cell carcinoma. Cancer. 2005 Nov 15;104(10):2084-91. doi: 10.1002/cncr.21470. PMID 16208700
- [Background] Dong H, Chen L. B7-H1 pathway and its role in the evasion of tumor immunity. J Mol Med (Berl). 2003 May;81(5):281-7. doi: 10.1007/s00109-003-0430-2. Epub 2003 Apr 30. PMID 12721664
- [Background] Azuma T, Yao S, Zhu G, Flies AS, Flies SJ, Chen L. B7-H1 is a ubiquitous antiapoptotic receptor on cancer cells. Blood. 2008 Apr 1;111(7):3635-43. doi: 10.1182/blood-2007-11-123141. Epub 2008 Jan 25. PMID 18223165
- [Background] Dong H, Strome SE, Salomao DR, Tamura H, Hirano F, Flies DB, Roche PC, Lu J, Zhu G, Tamada K, Lennon VA, Celis E, Chen L. Tumor-associated B7-H1 promotes T-cell apoptosis: a potential mechanism of immune evasion. Nat Med. 2002 Aug;8(8):793-800. doi: 10.1038/nm730. Epub 2002 Jun 24. PMID 12091876
- [Background] Iwai Y, Terawaki S, Honjo T. PD-1 blockade inhibits hematogenous spread of poorly immunogenic tumor cells by enhanced recruitment of effector T cells. Int Immunol. 2005 Feb;17(2):133-44. doi: 10.1093/intimm/dxh194. Epub 2004 Dec 20. PMID 15611321
- [Background] Iwai Y, Ishida M, Tanaka Y, Okazaki T, Honjo T, Minato N. Involvement of PD-L1 on tumor cells in the escape from host immune system and tumor immunotherapy by PD-L1 blockade. Proc Natl Acad Sci U S A. 2002 Sep 17;99(19):12293-7. doi: 10.1073/pnas.192461099. Epub 2002 Sep 6. PMID 12218188
- [Background] Strome SE, Dong H, Tamura H, Voss SG, Flies DB, Tamada K, Salomao D, Cheville J, Hirano F, Lin W, Kasperbauer JL, Ballman KV, Chen L. B7-H1 blockade augments adoptive T-cell immunotherapy for squamous cell carcinoma. Cancer Res. 2003 Oct 1;63(19):6501-5. PMID 14559843
- [Background] Hirano F, Kaneko K, Tamura H, Dong H, Wang S, Ichikawa M, Rietz C, Flies DB, Lau JS, Zhu G, Tamada K, Chen L. Blockade of B7-H1 and PD-1 by monoclonal antibodies potentiates cancer therapeutic immunity. Cancer Res. 2005 Feb 1;65(3):1089-96. PMID 15705911
- [Background] Blank C, Brown I, Peterson AC, Spiotto M, Iwai Y, Honjo T, Gajewski TF. PD-L1/B7H-1 inhibits the effector phase of tumor rejection by T cell receptor (TCR) transgenic CD8+ T cells. Cancer Res. 2004 Feb 1;64(3):1140-5. doi: 10.1158/0008-5472.can-03-3259. PMID 14871849
- [Background] Rizvi NA, Hellmann MD, Snyder A, Kvistborg P, Makarov V, Havel JJ, Lee W, Yuan J, Wong P, Ho TS, Miller ML, Rekhtman N, Moreira AL, Ibrahim F, Bruggeman C, Gasmi B, Zappasodi R, Maeda Y, Sander C, Garon EB, Merghoub T, Wolchok JD, Schumacher TN, Chan TA. Cancer immunology. Mutational landscape determines sensitivity to PD-1 blockade in non-small cell lung cancer. Science. 2015 Apr 3;348(6230):124-8. doi: 10.1126/science.aaa1348. Epub 2015 Mar 12. PMID 25765070
- [Background] Rizvi H, Sanchez-Vega F, La K, Chatila W, Jonsson P, Halpenny D, Plodkowski A, Long N, Sauter JL, Rekhtman N, Hollmann T, Schalper KA, Gainor JF, Shen R, Ni A, Arbour KC, Merghoub T, Wolchok J, Snyder A, Chaft JE, Kris MG, Rudin CM, Socci ND, Berger MF, Taylor BS, Zehir A, Solit DB, Arcila ME, Ladanyi M, Riely GJ, Schultz N, Hellmann MD. Molecular Determinants of Response to Anti-Programmed Cell Death (PD)-1 and Anti-Programmed Death-Ligand 1 (PD-L1) Blockade in Patients With Non-Small-Cell Lung Cancer Profiled With Targeted Next-Generation Sequencing. J Clin Oncol. 2018 Mar 1;36(7):633-641. doi: 10.1200/JCO.2017.75.3384. Epub 2018 Jan 16. PMID 29337640
- [Background] Hellmann MD, Nathanson T, Rizvi H, Creelan BC, Sanchez-Vega F, Ahuja A, Ni A, Novik JB, Mangarin LMB, Abu-Akeel M, Liu C, Sauter JL, Rekhtman N, Chang E, Callahan MK, Chaft JE, Voss MH, Tenet M, Li XM, Covello K, Renninger A, Vitazka P, Geese WJ, Borghaei H, Rudin CM, Antonia SJ, Swanton C, Hammerbacher J, Merghoub T, McGranahan N, Snyder A, Wolchok JD. Genomic Features of Response to Combination Immunotherapy in Patients with Advanced Non-Small-Cell Lung Cancer. Cancer Cell. 2018 May 14;33(5):843-852.e4. doi: 10.1016/j.ccell.2018.03.018. Epub 2018 Apr 12. PMID 29657128
- [Background] Hellmann MD, Ciuleanu TE, Pluzanski A, Lee JS, Otterson GA, Audigier-Valette C, Minenza E, Linardou H, Burgers S, Salman P, Borghaei H, Ramalingam SS, Brahmer J, Reck M, O'Byrne KJ, Geese WJ, Green G, Chang H, Szustakowski J, Bhagavatheeswaran P, Healey D, Fu Y, Nathan F, Paz-Ares L. Nivolumab plus Ipilimumab in Lung Cancer with a High Tumor Mutational Burden. N Engl J Med. 2018 May 31;378(22):2093-2104. doi: 10.1056/NEJMoa1801946. Epub 2018 Apr 16. PMID 29658845
- [Background] Hellmann MD, Rizvi NA, Goldman JW, Gettinger SN, Borghaei H, Brahmer JR, Ready NE, Gerber DE, Chow LQ, Juergens RA, Shepherd FA, Laurie SA, Geese WJ, Agrawal S, Young TC, Li X, Antonia SJ. Nivolumab plus ipilimumab as first-line treatment for advanced non-small-cell lung cancer (CheckMate 012): results of an open-label, phase 1, multicohort study. Lancet Oncol. 2017 Jan;18(1):31-41. doi: 10.1016/S1470-2045(16)30624-6. Epub 2016 Dec 5. PMID 27932067
- [Background] Beebe-Dimmer JL, Fryzek JP, Yee CL, Dalvi TB, Garabrant DH, Schwartz AG, Gadgeel S. Mesothelioma in the United States: a Surveillance, Epidemiology, and End Results (SEER)-Medicare investigation of treatment patterns and overall survival. Clin Epidemiol. 2016 Oct 26;8:743-750. doi: 10.2147/CLEP.S105396. eCollection 2016. PMID 27822122
- [Background] Vogelzang NJ, Rusthoven JJ, Symanowski J, Denham C, Kaukel E, Ruffie P, Gatzemeier U, Boyer M, Emri S, Manegold C, Niyikiza C, Paoletti P. Phase III study of pemetrexed in combination with cisplatin versus cisplatin alone in patients with malignant pleural mesothelioma. J Clin Oncol. 2003 Jul 15;21(14):2636-44. doi: 10.1200/JCO.2003.11.136. PMID 12860938
- [Background] Currie AJ, Prosser A, McDonnell A, Cleaver AL, Robinson BW, Freeman GJ, van der Most RG. Dual control of antitumor CD8 T cells through the programmed death-1/programmed death-ligand 1 pathway and immunosuppressive CD4 T cells: regulation and counterregulation. J Immunol. 2009 Dec 15;183(12):7898-908. doi: 10.4049/jimmunol.0901060. PMID 20007574
- [Background] Mansfield AS, Roden AC, Peikert T, Sheinin YM, Harrington SM, Krco CJ, Dong H, Kwon ED. B7-H1 expression in malignant pleural mesothelioma is associated with sarcomatoid histology and poor prognosis. J Thorac Oncol. 2014 Jul;9(7):1036-1040. doi: 10.1097/JTO.0000000000000177. PMID 24926549
- [Background] Alley EW, Lopez J, Santoro A, Morosky A, Saraf S, Piperdi B, van Brummelen E. Clinical safety and activity of pembrolizumab in patients with malignant pleural mesothelioma (KEYNOTE-028): preliminary results from a non-randomised, open-label, phase 1b trial. Lancet Oncol. 2017 May;18(5):623-630. doi: 10.1016/S1470-2045(17)30169-9. Epub 2017 Mar 11. PMID 28291584
- [Background] Gilligan D, Nicolson M, Smith I, Groen H, Dalesio O, Goldstraw P, Hatton M, Hopwood P, Manegold C, Schramel F, Smit H, van Meerbeeck J, Nankivell M, Parmar M, Pugh C, Stephens R. Preoperative chemotherapy in patients with resectable non-small cell lung cancer: results of the MRC LU22/NVALT 2/EORTC 08012 multicentre randomised trial and update of systematic review. Lancet. 2007 Jun 9;369(9577):1929-37. doi: 10.1016/S0140-6736(07)60714-4. PMID 17544497
- [Background] Brahmer JR, Drake CG, Wollner I, Powderly JD, Picus J, Sharfman WH, Stankevich E, Pons A, Salay TM, McMiller TL, Gilson MM, Wang C, Selby M, Taube JM, Anders R, Chen L, Korman AJ, Pardoll DM, Lowy I, Topalian SL. Phase I study of single-agent anti-programmed death-1 (MDX-1106) in refractory solid tumors: safety, clinical activity, pharmacodynamics, and immunologic correlates. J Clin Oncol. 2010 Jul 1;28(19):3167-75. doi: 10.1200/JCO.2009.26.7609. Epub 2010 Jun 1. PMID 20516446
- [Background] Eggermont AM, Chiarion-Sileni V, Grob JJ, Dummer R, Wolchok JD, Schmidt H, Hamid O, Robert C, Ascierto PA, Richards JM, Lebbe C, Ferraresi V, Smylie M, Weber JS, Maio M, Konto C, Hoos A, de Pril V, Gurunath RK, de Schaetzen G, Suciu S, Testori A. Adjuvant ipilimumab versus placebo after complete resection of high-risk stage III melanoma (EORTC 18071): a randomised, double-blind, phase 3 trial. Lancet Oncol. 2015 May;16(5):522-30. doi: 10.1016/S1470-2045(15)70122-1. Epub 2015 Mar 31. PMID 25840693
- [Background] Liu J, Blake SJ, Yong MC, Harjunpaa H, Ngiow SF, Takeda K, Young A, O'Donnell JS, Allen S, Smyth MJ, Teng MW. Improved Efficacy of Neoadjuvant Compared to Adjuvant Immunotherapy to Eradicate Metastatic Disease. Cancer Discov. 2016 Dec;6(12):1382-1399. doi: 10.1158/2159-8290.CD-16-0577. Epub 2016 Sep 23. PMID 27663893
- [Background] Forde PM, Chaft JE, Smith KN, Anagnostou V, Cottrell TR, Hellmann MD, Zahurak M, Yang SC, Jones DR, Broderick S, Battafarano RJ, Velez MJ, Rekhtman N, Olah Z, Naidoo J, Marrone KA, Verde F, Guo H, Zhang J, Caushi JX, Chan HY, Sidhom JW, Scharpf RB, White J, Gabrielson E, Wang H, Rosner GL, Rusch V, Wolchok JD, Merghoub T, Taube JM, Velculescu VE, Topalian SL, Brahmer JR, Pardoll DM. Neoadjuvant PD-1 Blockade in Resectable Lung Cancer. N Engl J Med. 2018 May 24;378(21):1976-1986. doi: 10.1056/NEJMoa1716078. Epub 2018 Apr 16. PMID 29658848
- [Background] Topalian SL, Hodi FS, Brahmer JR, Gettinger SN, Smith DC, McDermott DF, Powderly JD, Carvajal RD, Sosman JA, Atkins MB, Leming PD, Spigel DR, Antonia SJ, Horn L, Drake CG, Pardoll DM, Chen L, Sharfman WH, Anders RA, Taube JM, McMiller TL, Xu H, Korman AJ, Jure-Kunkel M, Agrawal S, McDonald D, Kollia GD, Gupta A, Wigginton JM, Sznol M. Safety, activity, and immune correlates of anti-PD-1 antibody in cancer. N Engl J Med. 2012 Jun 28;366(26):2443-54. doi: 10.1056/NEJMoa1200690. Epub 2012 Jun 2. PMID 22658127
- [Background] Carthon BC, Wolchok JD, Yuan J, Kamat A, Ng Tang DS, Sun J, Ku G, Troncoso P, Logothetis CJ, Allison JP, Sharma P. Preoperative CTLA-4 blockade: tolerability and immune monitoring in the setting of a presurgical clinical trial. Clin Cancer Res. 2010 May 15;16(10):2861-71. doi: 10.1158/1078-0432.CCR-10-0569. Epub 2010 May 11. PMID 20460488
- [Background] Woo SR, Turnis ME, Goldberg MV, Bankoti J, Selby M, Nirschl CJ, Bettini ML, Gravano DM, Vogel P, Liu CL, Tangsombatvisit S, Grosso JF, Netto G, Smeltzer MP, Chaux A, Utz PJ, Workman CJ, Pardoll DM, Korman AJ, Drake CG, Vignali DA. Immune inhibitory molecules LAG-3 and PD-1 synergistically regulate T-cell function to promote tumoral immune escape. Cancer Res. 2012 Feb 15;72(4):917-27. doi: 10.1158/0008-5472.CAN-11-1620. Epub 2011 Dec 20. PMID 22186141
- [Background] Chen H, Liakou CI, Kamat A, Pettaway C, Ward JF, Tang DN, Sun J, Jungbluth AA, Troncoso P, Logothetis C, Sharma P. Anti-CTLA-4 therapy results in higher CD4+ICOShi T cell frequency and IFN-gamma levels in both nonmalignant and malignant prostate tissues. Proc Natl Acad Sci U S A. 2009 Feb 24;106(8):2729-34. doi: 10.1073/pnas.0813175106. Epub 2009 Feb 6. PMID 19202079
- [Background] Liakou CI, Kamat A, Tang DN, Chen H, Sun J, Troncoso P, Logothetis C, Sharma P. CTLA-4 blockade increases IFNgamma-producing CD4+ICOShi cells to shift the ratio of effector to regulatory T cells in cancer patients. Proc Natl Acad Sci U S A. 2008 Sep 30;105(39):14987-92. doi: 10.1073/pnas.0806075105. Epub 2008 Sep 25. PMID 18818309
- [Background] Fu T, He Q, Sharma P. The ICOS/ICOSL pathway is required for optimal antitumor responses mediated by anti-CTLA-4 therapy. Cancer Res. 2011 Aug 15;71(16):5445-54. doi: 10.1158/0008-5472.CAN-11-1138. Epub 2011 Jun 27. PMID 21708958
- [Background] Borghaei H, Paz-Ares L, Horn L, Spigel DR, Steins M, Ready NE, Chow LQ, Vokes EE, Felip E, Holgado E, Barlesi F, Kohlhaufl M, Arrieta O, Burgio MA, Fayette J, Lena H, Poddubskaya E, Gerber DE, Gettinger SN, Rudin CM, Rizvi N, Crino L, Blumenschein GR Jr, Antonia SJ, Dorange C, Harbison CT, Graf Finckenstein F, Brahmer JR. Nivolumab versus Docetaxel in Advanced Nonsquamous Non-Small-Cell Lung Cancer. N Engl J Med. 2015 Oct 22;373(17):1627-39. doi: 10.1056/NEJMoa1507643. Epub 2015 Sep 27. PMID 26412456
- [Background] Schoenfeld J, Jinushi M, Nakazaki Y, Wiener D, Park J, Soiffer R, Neuberg D, Mihm M, Hodi FS, Dranoff G. Active immunotherapy induces antibody responses that target tumor angiogenesis. Cancer Res. 2010 Dec 15;70(24):10150-60. doi: 10.1158/0008-5472.CAN-10-1852. PMID 21159637
- [Background] Danilova L, Anagnostou V, Caushi JX, Sidhom JW, Guo H, Chan HY, Suri P, Tam A, Zhang J, Asmar ME, Marrone KA, Naidoo J, Brahmer JR, Forde PM, Baras AS, Cope L, Velculescu VE, Pardoll DM, Housseau F, Smith KN. The Mutation-Associated Neoantigen Functional Expansion of Specific T Cells (MANAFEST) Assay: A Sensitive Platform for Monitoring Antitumor Immunity. Cancer Immunol Res. 2018 Aug;6(8):888-899. doi: 10.1158/2326-6066.CIR-18-0129. Epub 2018 Jun 12. PMID 29895573
- [Background] Sivan A, Corrales L, Hubert N, Williams JB, Aquino-Michaels K, Earley ZM, Benyamin FW, Lei YM, Jabri B, Alegre ML, Chang EB, Gajewski TF. Commensal Bifidobacterium promotes antitumor immunity and facilitates anti-PD-L1 efficacy. Science. 2015 Nov 27;350(6264):1084-9. doi: 10.1126/science.aac4255. Epub 2015 Nov 5. PMID 26541606
- [Background] Noone AM, Howlader N, Krapcho M, et al. SEER cancer statistics review, 1975-2015, National Cancer institute, Bethesda, MD, 2018.
- [Background] Quispel-Janssen J, Zago G, Schouten R, et al. OA13.01 A phase II study of nivolumab in malignant pleural mesothelioma (NivoMes): With translational research (TR) biopsies. J Thorac Oncol. 2017;12(1):s293.
- [Background] Baas P, Disselhorst MJ, Harms E, et al. PL02.04: Ipilimumab and nivolumab in the treatment of malignant pleural mesothelioma: Final results of a phase II study (initiate). 14th International Conference of the International Mesothelioma Interest Group. 2018.
- [Background] Scherpereel A, Mazieres J, Greillier L, et al. Second- or third-line nivolumab (nivo) versus nivo plus ipilimumab (ipi) in malignant pleural mesothelioma (MPM) patients: Results of the IFCT-1501 MAPS2 randomized phase II trial. JCO. 2017;35(18):LBA8507.
- [Background] de Perrot M, Feld R, Cho BC, Bezjak A, Anraku M, Burkes R, Roberts H, Tsao MS, Leighl N, Keshavjee S, Johnston MR. Trimodality therapy with induction chemotherapy followed by extrapleural pneumonectomy and adjuvant high-dose hemithoracic radiation for malignant pleural mesothelioma. J Clin Oncol. 2009 Mar 20;27(9):1413-8. doi: 10.1200/JCO.2008.17.5604. Epub 2009 Feb 17. PMID 19224855
- [Background] Sabatino M, Kim-Schulze S, Panelli MC, Stroncek D, Wang E, Taback B, Kim DW, Deraffele G, Pos Z, Marincola FM, Kaufman HL. Serum vascular endothelial growth factor and fibronectin predict clinical response to high-dose interleukin-2 therapy. J Clin Oncol. 2009 Jun 1;27(16):2645-52. doi: 10.1200/JCO.2008.19.1106. Epub 2009 Apr 13. PMID 19364969
- [Background] Blazar BR, Carreno BM, Panoskaltsis-Mortari A, Carter L, Iwai Y, Yagita H, Nishimura H, Taylor PA. Blockade of programmed death-1 engagement accelerates graft-versus-host disease lethality by an IFN-gamma-dependent mechanism. J Immunol. 2003 Aug 1;171(3):1272-7. doi: 10.4049/jimmunol.171.3.1272. PMID 12874215
- [Background] Zalcman G, Mazieres J, Margery J, Greillier L, Audigier-Valette C, Moro-Sibilot D, Molinier O, Corre R, Monnet I, Gounant V, Riviere F, Janicot H, Gervais R, Locher C, Milleron B, Tran Q, Lebitasy MP, Morin F, Creveuil C, Parienti JJ, Scherpereel A; French Cooperative Thoracic Intergroup (IFCT). Bevacizumab for newly diagnosed pleural mesothelioma in the Mesothelioma Avastin Cisplatin Pemetrexed Study (MAPS): a randomised, controlled, open-label, phase 3 trial. Lancet. 2016 Apr 2;387(10026):1405-1414. doi: 10.1016/S0140-6736(15)01238-6. Epub 2015 Dec 21. PMID 26719230
- [Background] Scagliotti G, Gaafar R, Nowak A, et al. PL02.09 nintedanib + pemetrexed/cisplatin in patients with unresectable MPM: Phase III results from the lume-meso trial. IASLC 19th World Conference on Lung Cancer.
- [Background] Thapa B, Salcedo A, Lin X, Walkiewicz M, Murone C, Ameratunga M, Asadi K, Deb S, Barnett SA, Knight S, Mitchell P, Watkins DN, Boutros PC, John T. The Immune Microenvironment, Genome-wide Copy Number Aberrations, and Survival in Mesothelioma. J Thorac Oncol. 2017 May;12(5):850-859. doi: 10.1016/j.jtho.2017.02.013. Epub 2017 Feb 28. PMID 28257959
- [Background] Desai A, Karrison T, Rose B, et al. OA08.03 phase II trial of pembrolizumab (NCT02399371) in previously treated malignant mesothelioma: Final analysis. J Thorac Oncol. 2018;13(10):S339.
- [Background] Nakano T, Okada M, Kijima T, et al. OA08.01 long-term efficacy and safety of nivolumab in second- or third-line japanese malignant pleural mesothelioma patients (phase II: MERIT study). J Thorac Oncol. 2018;13(10):S338.
- [Background] Nowak AK, Sei Kok P, Joost Lesterhuis W, et al. OA08.02 DREAM - A phase 2 trial of durvalumab with first line chemotherapy in mesothelioma: Final result. J Thorac Oncol. 2018;13(10):S339.
- [Background] Rozeman EA, Blank CU, Van Akkooi A,Christopher Jonathan, et al. Neoadjuvant ipilimumab + nivolumab (IPI+NIVO) in palpable stage III melanoma: Updated data from the OpACIN trial and first immunological analyses. JCO. 2017;35(15):9586.
- [Background] Schmid P, Park YH, Muñoz-Couselo E, et al. Pembrolizumab (pembro) + chemotherapy (chemo) as neoadjuvant treatment for triple negative breast cancer (TNBC): Preliminary results from KEYNOTE-173. JCO. 2017;35(15):556.
- [Background] Nanda R, Liu MC, Yau C, et al. Pembrolizumab plus standard neoadjuvant therapy for high-risk breast cancer (BC): Results from I-SPY 2. JCO. 2017;35(15):506.
- [Background] Directive 2001/20/EC of the european parliament and of the council of 4 april 2001. Official Journal of the European Communities. 2001;L(121):35,36,37,38,39,40,41,42,43,44.
- [Background] Powderly JD, Koeppen H, Hodi FS, et al. Biomarkers and associations with the clinical activity of PD-L1 blockade in a MPDL3280A study. JCO. 2013;31(15):3001.
- [Background] Vetizou M, Pitt JM, Daillere R, Lepage P, Waldschmitt N, Flament C, Rusakiewicz S, Routy B, Roberti MP, Duong CP, Poirier-Colame V, Roux A, Becharef S, Formenti S, Golden E, Cording S, Eberl G, Schlitzer A, Ginhoux F, Mani S, Yamazaki T, Jacquelot N, Enot DP, Berard M, Nigou J, Opolon P, Eggermont A, Woerther PL, Chachaty E, Chaput N, Robert C, Mateus C, Kroemer G, Raoult D, Boneca IG, Carbonnel F, Chamaillard M, Zitvogel L. Anticancer immunotherapy by CTLA-4 blockade relies on the gut microbiota. Science. 2015 Nov 27;350(6264):1079-84. doi: 10.1126/science.aad1329. Epub 2015 Nov 5. PMID 26541610
- [Derived] Reuss JE, Lee PK, Mehran RJ, Hu C, Ke S, Jamali A, Najjar M, Niknafs N, Wehr J, Oner E, Meng Q, Pereira G, Hosseini-Nami S, Sausen M, Zahurak M, Battafarano RJ, Hales RK, Friedberg J, Sepesi B, Deutsch JS, Cottrell T, Taube J, Illei PB, Smith KN, Pardoll DM, Tsao AS, Brahmer JR, Anagnostou V, Forde PM. Perioperative nivolumab or nivolumab plus ipilimumab in resectable diffuse pleural mesothelioma: a phase 2 trial and ctDNA analyses. Nat Med. 2025 Dec;31(12):4097-4108. doi: 10.1038/s41591-025-03958-3. Epub 2025 Sep 8. PMID 40921804